CLINICAL TRIAL: NCT00579904
Title: Walnuts, Walnut-Oil, Glucose Homeostasis, PCOS
Brief Title: The Effects of Walnuts, Walnut-Oil, Almonds and Fish Oils on Glucose Homeostasis in Polycystic Ovary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200513651; R21AT002280 (NIH)
Record Dates: First submitted 2007-12-17; First posted 2007-12-24 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2016-10

CONDITIONS: Polycystic Ovary Syndrome; Insulin Resistance
Keywords: PCOS; polycystic ovary syndrome; insulin resistance; fish oil; walnut-oil; walnuts; almonds; monounsaturated fats; polyunsaturated fats; MUFA; PUFA
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- walnuts (Active Comparator): Patients will be randomized to receive walnuts
  Interventions: Dietary Supplement: walnuts
- almonds (Active Comparator): Patients will be randomized to receive almonds
  Interventions: Dietary Supplement: almonds

INTERVENTIONS:
Dietary Supplement: walnuts — Subjects will follow their usual diet for 4 weeks; after that they will be randomized to walnuts. They will eat walnuts once daily for six weeks.
  Arms: walnuts
Dietary Supplement: almonds — Subjects will follow their usual diet for 4 weeks; after that they will be randomized to almonds. They will eat almonds once daily for six weeks.
  Arms: almonds

SUMMARY:
The purpose of this study is to learn more about the effects of walnuts, walnut-oil, almonds and fish oils on blood sugar and insulin levels in polycystic ovary syndrome (PCOS) patients. The hypothesis is that a diet rich in these foods will improve insulin resistance in women with PCOS.

DETAILED DESCRIPTION:
Polycystic ovary syndrome is a common disease that affects 1 out of 16 women. Metabolic and endocrine abnormalities seen in PCOS include insulin resistance, androgen excess and infertility. This study focuses on the insulin resistance aspect because increased insulin resistance leads to premature onset of impaired glucose tolerance or diabetes whereas decreased insulin resistance reduces androgen excess, improves the ovarian function and increases fertility. Although insulin resistance can be treated with insulin-sensitizing drugs, PCOS clinically manifests during adolescence and the long-term safety of the drug-treatment can be a concern. Thus, improving insulin resistance with effective nutritional approaches would be very desirable. Epidemiological studies and animal experiments suggest that replacement of dietary saturated fats with monounsaturated (MUFA) and polyunsaturated (PUFA) fats improves insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of polycystic ovary syndrome
* Body mass index (BMI) 22-52

Exclusion Criteria:

* Habitual dietary intake of less than 30% fat
* Use of oral contraceptives, insulin sensitizers, d-chiro inositol, or any other supplements affecting weight or insulin sensitivity during the preceding two months
* Impaired glucose tolerance
* Diabetes mellitus
* Other system illnesses such as renal, hepatic, gastrointestinal, severe hyperlipidemia and hypertension that require medication
* Smoking, alcohol intake (more than 2 drinks/week)
* The laboratory values used for exclusion of subjects will be fasting glucose > 110 mg/dl, glycosylated hemoglobin (HgBA1) > 6.5%, serum creatinine > 1.5 mg/dl, ALT or AST > 2x the upper limit of normal, cholesterol > 250 mg/dl. The investigators will also exclude subjects with hematocrit < 30%.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2006-04; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
The investigators hope to learn the effects of walnuts, walnut-oil, almonds and fish oils on blood sugar and insulin levels in PCOS patients. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Sidika E Kasim-Karakas, MD, Principal Investigator — University of California, Davis
Locations (1):
- Clinical and Translational Science Center Clinical Resources Center (CCRC), Mather, California, United States

IPD SHARING:
Plan to Share IPD: No